CLINICAL TRIAL: NCT00159874
Title: A Multicenter, Long-Term Extension Study to Assess Safety of Oral Sildenafil Citrate In The Treatment Of Subjects Who Have Completed Study A1481131
Brief Title: A Long Term Extension Study Evaluating Safety Of Sildenafil Citrate When Used To Treat Pulmonary Arterial Hypertension (PAH) In Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A1481156
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: children
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sildenafil high dose (Experimental): As per Protocol Amendment 8 (Aug 2011), all doses in the high dose treatment group were discontinued. Subjects who were receiving these doses and continued in the study were requested to down titrate.
  Interventions: Drug: Sildenafil citrate
- Sildenafil Low dose (Experimental)
  Interventions: Drug: Sildenafil citrate
- Sildenafil medium dose (Experimental): As per Protocol Amendment 8 (August 2011), the dose 40 mg TID in the medium dose treatment group was discontinued. Subjects who were receiving this dose and continued in the study were requested to down titrate.
  Interventions: Drug: Sildenafil citrate

INTERVENTIONS:
Drug: Sildenafil citrate — Oral, subjects with body weight ≥8 - 20 kg: 20 mg 3 times a day (tid) subjects with body weight >20 - 45 kg: 40 mg 3 times a day (tid) subjects with body weight >45 kg: 80 mg 3 times a day (tid)
  Arms: Sildenafil high dose
Drug: Sildenafil citrate — Oral,10 mg 3 times a day (tid), only subjects with body weight >20 kg
  Arms: Sildenafil Low dose
Drug: Sildenafil citrate — Oral, subjects with body weight ≥8 - 20 kg: 10 mg 3 times a day (tid); subjects with body weight >20 - 45 kg: 20 mg 3 times a day (tid); subjects with body weight >45 kg: 40 mg 3 times a day (tid)
  Arms: Sildenafil medium dose

SUMMARY:
Active treatment, dose-blinded extension study evaluating the safety and long term efficacy of sildenafil citrate in children with PAH.

ELIGIBILITY:
Inclusion Criteria:

* Patients must complete the 16 Week double-blind efficacy study A1481131.

Exclusion Criteria:

* Any patient who did not complete Study A1481131.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 234 (Actual)
Dates: Start 2004-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (31):
- United States (10):
  - Pfizer Investigational Site, Palo Alto, California
  - Pfizer Investigational Site, Stanford, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Seattle, Washington
- Pfizer Investigational Site, São Paulo, São Paulo, Brazil
- Pfizer Investigational Site, Puente Alto, Santiago Metropolitan, Chile
- Colombia (2):
  - Pfizer Investigational Site, Medellín, Antioquia
  - Pfizer Investigational Site, Bogota, Cundinamarca
- Pfizer Investigational Site, Guatemala City, Guatemala
- Hungary (2):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Szeged
- India (2):
  - Pfizer Investigational Site, Hyderabad, Andhra Pradesh
  - Pfizer Investigational Site, Kochi, Kerala
- Pfizer Investigational Site, Bologna, Italy
- Pfizer Investigational Site, Tokyo, Japan
- Pfizer Investigational Site, George Town, Pulau Pinang, Malaysia
- Pfizer Investigational Site, Mexico City, Mexico City, Mexico
- Poland (4):
  - Pfizer Investigational Site, Krakow
  - Pfizer Investigational Site, Ruda Śląska
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Zabrze
- Pfizer Investigational Site, Moscow, Russia
- Pfizer Investigational Site, Lund, Sweden
- Taiwan (2):
  - Pfizer Investigational Site, Kaohsiung City
  - Pfizer Investigational Site, Taipei

REFERENCES:
- [Derived] Russell S, Beghetti M, Oudiz R, Balagtas C, Zhang M, Ivy D. Effects of oral sildenafil on exercise capacity in children with pulmonary arterial hypertension: a randomised trial. Open Heart. 2019 Dec 3;6(2):e001149. doi: 10.1136/openhrt-2019-001149. eCollection 2019. PMID 31908813
- [Derived] Chanu P, Gao X, Bruno R, Claret L, Harnisch L. A modeling and simulation-based assessment of the impact of confounding factors on the readout of a sildenafil survival trial in pulmonary arterial hypertension. J Pharmacokinet Pharmacodyn. 2019 Oct;46(5):499-509. doi: 10.1007/s10928-019-09654-3. Epub 2019 Sep 20. PMID 31538282
- [Derived] Barst RJ, Beghetti M, Pulido T, Layton G, Konourina I, Zhang M, Ivy DD; STARTS-2 Investigators. STARTS-2: long-term survival with oral sildenafil monotherapy in treatment-naive pediatric pulmonary arterial hypertension. Circulation. 2014 May 13;129(19):1914-23. doi: 10.1161/CIRCULATIONAHA.113.005698. Epub 2014 Mar 17. PMID 24637559
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481156&StudyName=A%20Long%20Term%20Extension%20Study%20Evaluating%20Safety%20Of%20Sildenafil%20Citrate%20When%20Used%20To%20Treat%20Pulmonary%20Arterial%20Hypertension%20%28PAH%29%20In%20Chil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This extension study included 220 participants at 31 sites. 14 participants did not go from A1481131 (NCT00159913) to A1481156. Participants from one center in Canada participated in base study A1481131 (NCT00159913) but not in this extension study.
Pre-assignment Details: Participants remained in the same dose group as in study A1481131 (NCT00159913). Participants randomized to placebo in NCT00159913 were rerandomized to sildenafil in A1481156. Placebo participants in low weight category were rerandomized to medium or high dose (1:2) and other weight categories were rerandomized to low, medium or high dose (1:1:1).
Groups:
- Sildenafil Low/Low Dose: Participants randomized to sildenafil low dose in study A1481131 (NCT00159913) and in the extension study A1481156
- Sildenafil Medium/ Medium Dose: Participants randomized to sildenafil medium dose in study A1481131 (NCT00159913) and in the extension study A1481156
- Sildenafil High/ High Dose: Participants randomized to sildenafil high dose in study A1481131 (NCT00159913) and in the extension study A1481156
- Placebo/ Low Dose: Participants randomized to placebo in study A1481131 (NCT00159913) and randomized to sildenafil low dose in study A1481156
- Placebo/ Medium Dose: Participants randomized to placebo in study A1481131 (NCT00159913) and randomized to sildenafil medium dose in study A1481156
- Placebo/ High Dose: Participants randomized to placebo in study A1481131 (NCT00159913) and randomized to sildenafil high dose in study A1481156
- Placebo Non-randomized: This group comprised those placebo participants who either discontinued from base study A1481131 (NCT00159913) or chose not to enter study A1481156 and hence not randomly assigned to a sildenafil dose group at the start of study A1481156
Period: Overall Study
Arm/Group | Sildenafil Low/Low Dose | Sildenafil Medium/ Medium Dose | Sildenafil High/ High Dose | Placebo/ Low Dose | Placebo/ Medium Dose | Placebo/ High Dose | Placebo Non-randomized
Started | 42 | 55 | 77 | 13 | 19 | 23 | 5
Treated | 42 | 55 | 77 | 13 | 19 | 23 | 5
Completed | 22 | 25 | 34 | 7 | 11 | 11 | 0
Not Completed | 20 | 30 | 43 | 6 | 8 | 12 | 5
Not completed — Adverse Event | 2 | 2 | 5 | 1 | 1 | 2 | 0
Not completed — Does Not Meet Entrance Criteria | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 1 | 1 | 0 | 3 | 0
Not completed — Lost to Follow-up | 1 | 0 | 3 | 0 | 1 | 2 | 1
Not completed — Other | 8 | 8 | 8 | 0 | 2 | 1 | 3
Not completed — Protocol Violation | 0 | 5 | 2 | 0 | 0 | 0 | 0
Not completed — Death | 3 | 8 | 15 | 0 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 6 | 8 | 4 | 3 | 2 | 1
Not completed — Pregnancy | 1 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sildenafil Low/Low Dose | Sildenafil Medium/ Medium Dose | Sildenafil High/ High Dose | Placebo/ Low Dose | Placebo/ Medium Dose | Placebo/ High Dose | Placebo Non-randomized | Total
Number analyzed (Participants) | 42 | 55 | 77 | 13 | 19 | 23 | 5 | 234
Age, Customized [Number; unit: Participants]
  1-4 | 0 | 9 | 19 | 1 | 3 | 2 | 1 | 35
  5-12 | 25 | 28 | 36 | 11 | 10 | 14 | 2 | 126
  13-17 | 17 | 18 | 22 | 1 | 6 | 7 | 2 | 73
  >=18 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 31 | 51 | 9 | 11 | 15 | 3 | 145
  Male | 17 | 24 | 26 | 4 | 8 | 8 | 2 | 89

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting at Least One Adverse Event
Description: Safety was measured according to standard adverse event collection as described in the adverse event section of the results. Complete tables of the adverse events according to the A1481156 treatment groups are provided in the reported adverse event section.
Time Frame: Up to Follow-Up visit (30 to 40 days after study completion or treatment discontinuation)
Population: The safety population consisted of all participants who had taken at least one dose of study medication in A1481131 (NCT00159913).
Measure: Number; unit: Participants
Arm/Group | Sildenafil Low/Low Dose | Sildenafil Medium/ Medium Dose | Sildenafil High/ High Dose | Placebo/ Low Dose | Placebo/ Medium Dose | Placebo/ High Dose | Placebo Non-randomized
Number analyzed (Participants) | 42 | 55 | 77 | 13 | 19 | 23 | 5
Participants | 41 | 55 | 73 | 13 | 19 | 22 | 3

2. Primary Outcome: Number of Participants Reporting Treatment-related Adverse Events
Description: Safety was measured according to standard adverse event collection as described in the adverse event section of the results.
Time Frame: Up to Follow-Up visit (30 to 40 days after study completion or treatment discontinuation)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Sildenafil Low/Low Dose | Sildenafil Medium/ Medium Dose | Sildenafil High/ High Dose | Placebo/ Low Dose | Placebo/ Medium Dose | Placebo/ High Dose | Placebo Non-randomized
Number analyzed (Participants) | 42 | 55 | 77 | 13 | 19 | 23 | 5
Participants | 20 | 24 | 41 | 9 | 9 | 11 | 3

3. Primary Outcome: Number of Participants Reporting at Least One Serious Adverse Event
Description: Safety was measured according to standard adverse event collection as described in the adverse event section of the results. Complete tables of the serious adverse events according to the A1481156 treatment groups are provided in the reported adverse event section.
Time Frame: Up to Follow-Up visit (30 to 40 days after study completion or treatment discontinuation)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Sildenafil Low/Low Dose | Sildenafil Medium/ Medium Dose | Sildenafil High/ High Dose | Placebo/ Low Dose | Placebo/ Medium Dose | Placebo/ High Dose | Placebo Non-randomized
Number analyzed (Participants) | 42 | 55 | 77 | 13 | 19 | 23 | 5
Participants | 13 | 33 | 38 | 1 | 4 | 10 | 0

4. Primary Outcome: Number of Participants Reporting Treatment-related Serious Adverse Events
Description: All serious adverse events regardless of treatment group or suspected relationship to study drug were reported. Investigators were to provide independent determination of possible causality of any serious adverse event.
Time Frame: Up to Follow-Up visit (30 to 40 days after study completion or treatment discontinuation)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Sildenafil Low/Low Dose | Sildenafil Medium/ Medium Dose | Sildenafil High/ High Dose | Placebo/ Low Dose | Placebo/ Medium Dose | Placebo/ High Dose | Placebo Non-randomized
Number analyzed (Participants) | 42 | 55 | 77 | 13 | 19 | 23 | 5
Participants | 1 | 1 | 4 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Deaths Reported in the Study Prior to the Data Monitoring Committee (DMC) Recommendation of Dose Down Titration
Description: Deaths were reported immediately independent of the circumstances or suspected cause at any time during the study through the last follow-up visit or 30 days after the last administration of study drug, whichever comes later.
Time Frame: Pre-DMC Recommendation dose down titration (04 August 2011)
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- Sildenafil Low Dose: Participants randomized to sildenafil low dose in study A1481131 (NCT00159913) and continued in the low dose group in the extension study A1481156, and participants randomized to placebo dose in study A1481131 (NCT00159913) and randomized to sildenafil low dose in the extension study A1481156
- Sildenafil Medium Dose: Participants randomized to sildenafil medium dose in study A1481131 (NCT00159913) and continued in the medium dose group in the extension study A1481156, and participants randomized to placebo dose in study A1481131 (NCT00159913) and randomized to sildenafil medium dose in the extension study A1481156
- Sildenafil High Dose: Participants randomized to sildenafil high dose in study A1481131 (NCT00159913)and continued in the high dose group in the extension study A1481156, and participants randomized to placebo dose in study A1481131 (NCT00159913) and randomized to sildenafil high dose in the extension study A1481156
Arm/Group | Sildenafil Low Dose | Sildenafil Medium Dose | Sildenafil High Dose
Number analyzed (Participants) | 55 | 74 | 100
Participants | 5 | 10 | 22

6. Primary Outcome: Number of Deaths Reported During This Study
Description: as for outcome 5
Time Frame: Last follow-up visit or 30 days after the last administration of study drug
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- Sildenafil Low Dose: Participants randomized to sildenafil low dose in study A1481131 (NCT00159913)and continued in the low dose group in the extension study A1481156, and participants randomized to placebo dose in study A1481131 (NCT00159913) and randomized to sildenafil low dose in the extension study A1481156
Arm/Group | Sildenafil Low Dose | Sildenafil Medium Dose | Sildenafil High Dose
Number analyzed (Participants) | 55 | 74 | 100
Participants | 5 | 13 | 24

7. Primary Outcome: Discontinuation Due to Intolerability
Description: Participant who experienced drug-related intolerance, the participant's dose was reduced by 50%. If, after a dose reduction, the participant continued to appear intolerant, they were discontinued from study treatment.
Time Frame: Throughout the treatment duration (median treatment duration 1689 to 1744 days)
Population: Safety population included all randomly assigned participants who took at least 1 dose of study medication in Study A1481131 (NCT00159913).
Measure: Number; unit: Participants
Arm/Group | Sildenafil Low Dose | Sildenafil Medium Dose | Sildenafil High Dose
Number analyzed (Participants) | 55 | 74 | 100
Participants | 2 | 1 | 3

8. Primary Outcome: Downtitration in Dose Due to Intolerability.
Description: Based on review of the survival data, DMC concluded that the high dose of sildenafil was associated with a harmful effect on survival when compared to the low dose. The DMC also expressed concern as to the potential dose-response relationship between increasing dose and mortality. Therefore, on 04 August 2011, the DMC recommended discontinuation of the 40 mg and 80 mg three times a day (TID) doses, as well as the 20 mg TID dose in children with body weight ≤20 kg. The protocol was amended per DMC recommendations.
Time Frame: Pre-DMC recomendation (04 August 2011)
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | Sildenafil Low/Low Dose | Sildenafil Medium/ Medium Dose | Sildenafil High/ High Dose | Placebo/ Low Dose | Placebo/ Medium Dose | Placebo/ High Dose | Placebo Non-randomized
Number analyzed (Participants) | 42 | 55 | 77 | 13 | 19 | 23 | 5
Participants | 0 | 0 | 3 | 0 | 2 | 1 | 0

9. Primary Outcome: Number of Participants With Deterioration Post Baseline in Visual Acuity Safety Tests
Description: Visual Acuity is measured either using the reduced Snellen test or via Teller cards, and was assessed in the left and right eyes separately. There were 9 lines on the reduced Snellen chart which were coded as 6/60, 6/36, 6/24, 6/18, 6/12, 6/9, 6/6, 6/5, 6/4 (where 6/60 was the easiest to read and 6/4 was the most difficult to read). If a participant experienced a visual adverse event the investigator was asked to perform additional ocular assessments either at the visit when the participant reported the visual adverse event or at an unplanned visit.
Time Frame: Week 36
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | Sildenafil Low/Low Dose | Sildenafil Medium/ Medium Dose | Sildenafil High/ High Dose | Placebo/ Low Dose | Placebo/ Medium Dose | Placebo/ High Dose | Placebo Non-randomized
Number analyzed (Participants) | 42 | 55 | 77 | 13 | 19 | 23 | 5
Participants | 10 | 11 | 17 | 0 | 4 | 4 | 0

10. Primary Outcome: Number of Participants With Deterioration Post Baseline in Color Vision Monitoring Safety Tests.
Description: Colour vision was measured where appropriate via the Farnsworth-Munsell D-15 Hue test. This test was performed in both eyes simultaneously or just in a single specific eye. If using a single eye the same eye was used throughout the study. In case of young participants an age-and-ability-appropriate evaluation such as the Ishihara Test for Unlettered Persons were conducted.
Time Frame: Week 36
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | Sildenafil Low/Low Dose | Sildenafil Medium/ Medium Dose | Sildenafil High/ High Dose | Placebo/ Low Dose | Placebo/ Medium Dose | Placebo/ High Dose | Placebo Non-randomized
Number analyzed (Participants) | 42 | 55 | 77 | 13 | 19 | 23 | 5
Participants | 2 | 2 | 1 | 0 | 0 | 1 | 1

11. Primary Outcome: Pediatric Cognitive Development Status at Week 16.
Description: Participant's cognitive development status was assessed at A1481156 baseline (Week 16 in A1481131; NCT00159913) using the physician assessment questions. Assessment question (i.e., compared to other children the participant's age group is this participant's cognitive development limited?) included the following criteria : severely limited, moderately limited, mildly limited and not limited.
Time Frame: Week 16
Population: Safety population included all randomly assigned participants who took at least 1 dose of study medication in Study A1481131 (NCT00159913). Participants with observed data were included in table.
Measure: Number; unit: Participants
Arm/Group | Sildenafil Low/Low Dose | Sildenafil Medium/ Medium Dose | Sildenafil High/ High Dose | Placebo/ Low Dose | Placebo/ Medium Dose | Placebo/ High Dose | Placebo Non-randomized
Number analyzed (Participants) | 42 | 55 | 77 | 13 | 19 | 23 | 5
Participants
  Severely Limited | 2 | 4 | 2 | 0 | 1 | 1 | 0
  Moderately Limited | 5 | 6 | 8 | 1 | 5 | 2 | 1
  Mildly Limited | 6 | 7 | 12 | 1 | 1 | 1 | 0
  Not Limited | 26 | 38 | 54 | 11 | 12 | 19 | 1

12. Primary Outcome: Pediatric Cognitive Development Status at Week 52.
Description: Participant's cognitive development status was assessed at Week 52 using the physician assessment questions. Assessment question (i.e., compared to other children the participant's age group is this participant's cognitive development limited?) included the following criteria : severely limited, moderately limited, mildly limited and not limited.
Time Frame: Week 52
Population: as for outcome 11
Measure: Number; unit: Participants
Arm/Group | Sildenafil Low/Low Dose | Sildenafil Medium/ Medium Dose | Sildenafil High/ High Dose | Placebo/ Low Dose | Placebo/ Medium Dose | Placebo/ High Dose
Number analyzed (Participants) | 42 | 55 | 77 | 13 | 19 | 23
Participants
  Severely Limited | 1 | 1 | 2 | 0 | 0 | 0
  Moderately Limited | 5 | 10 | 6 | 1 | 5 | 2
  Mildly Limited | 3 | 5 | 8 | 0 | 3 | 3
  Not Limited | 27 | 36 | 50 | 11 | 10 | 15

13. Primary Outcome: Pediatric Motor Development Status at Week 16.
Description: Participant's motor development status was assessed at A1481156 baseline (Week 16 in A1481131; NCT00159913) using the physician assessment questions. Assessment question (i.e., compared to other children the participant's age group is this participant's motor development limited?) included the following criteria : severely limited, moderately limited, mildly limited and not limited.
Time Frame: Week 16
Population: as for outcome 11
Measure: Number; unit: Participants
Arm/Group | Sildenafil Low/Low Dose | Sildenafil Medium/ Medium Dose | Sildenafil High/ High Dose | Placebo/ Low Dose | Placebo/ Medium Dose | Placebo/ High Dose | Placebo Non-randomized
Number analyzed (Participants) | 42 | 55 | 77 | 13 | 19 | 23 | 5
Participants
  Severely Limited | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Moderately Limited | 5 | 5 | 7 | 0 | 4 | 1 | 1
  Mildly Limited | 10 | 11 | 20 | 1 | 5 | 2 | 0
  Not Limited | 24 | 39 | 49 | 12 | 9 | 20 | 1

14. Primary Outcome: Pediatric Motor Development Status at Week 52
Description: Participant's motor development status was assessed at Week 52 using the physician assessment questions. Assessment question (i.e., compared to other children the participant's age group is this participant's motor development limited?) included the following criteria : severely limited, moderately limited, mildly limited and not limited.
Time Frame: Week 52
Population: as for outcome 11
Measure: Number; unit: Participants
Arm/Group | Sildenafil Low/Low Dose | Sildenafil Medium/ Medium Dose | Sildenafil High/ High Dose | Placebo/ Low Dose | Placebo/ Medium Dose | Placebo/ High Dose
Number analyzed (Participants) | 42 | 55 | 77 | 13 | 19 | 23
Participants
  Severely Limited | 0 | 0 | 0 | 0 | 0 | 0
  Moderately Limited | 4 | 9 | 5 | 0 | 2 | 0
  Mildly Limited | 8 | 8 | 15 | 3 | 6 | 3
  Not Limited | 24 | 35 | 46 | 9 | 10 | 17

15. Secondary Outcome: Peak Volume of Oxygen (VO2) Consumed at Year 1 Using a Bicycle Ergometry Cardiopulmonary Exercise Test (CPX)
Description: Exercise Tolerance Test (CPX test) was performed on developmentally able participants to determine the peak volume of VO2 consumed. Participants were assumed to be developmentally able if they had a CPX exercise assessment at any visit during study A1481131 (NCT00159913). The CPX tests were performed as close to trough plasma levels of sildenafil as possible, i.e., prior to dosing and at least 4 hours after the previous dose. If participants were able to perform the CPX test in Study A1481131 (NCT00159913), they were expected to be able to perform the exercise paradigm in the extension study (A1481156) unless their clinical condition had deteriorated and the investigator considered this was unsafe for the participant
Time Frame: 1 year
Population: An ITT population included all randomized participants who took at least 1 dose of study medication in base study and certain analyses were conducted at pre-specified time points: 1, 2 years and 3, 4 and 5 years (where data quantity allowed) from A1481131 (NCT00159913) baseline. Only developmentally able participants were used for this analysis.
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | Sildenafil Low Dose | Sildenafil Medium Dose | Sildenafil High Dose
Number analyzed (Participants) | 38 | 36 | 40
mL/kg/min | 19.97 (5.17) | 18.69 (5.92) | 17.93 (4.02)
Statistical Analysis 1: Comparison: Sildenafil Low Dose vs Sildenafil Medium Dose; Analyses were performed using analysis of covariance with etiology, weight, day of assessment and baseline peak VO2 as the covariates; Test type: Superiority or Other; p = 0.253, ANCOVA; Least Square Mean Difference = -7.02, 95% CI 2-sided [-19.13 to 5.09], Standard Error of Mean 6.10 — Least square mean difference of -7.02 was calculated as ' Sildenafil Medium Dose - Low Dose'
Statistical Analysis 2: Comparison: Sildenafil Low Dose vs Sildenafil High Dose; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p = 0.100, ANCOVA; Least Square Mean Difference = -9.84, 95% CI 2-sided [-21.60 to 1.93], Standard Error of Mean 5.92 — Least square mean difference of -9.84 was calculated as ' Sildenafil High Dose - Low Dose'
Statistical Analysis 3: Comparison: Sildenafil Medium Dose vs Sildenafil High Dose; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p = 0.640, ANCOVA; Least Square Mean Difference = -2.82, 95% CI 2-sided [-14.75 to 9.11], Standard Error of Mean 6.01 — Least square mean difference of -2.82 was calculated as ' Sildenafil High Dose - Medium Dose'

16. Secondary Outcome: Percentage Change From Baseline in Percent Predicted Peak VO2 at Year 1.
Description: Exercise Tolerance Test (CPX test) was performed on developmentally able participants to measure the percent predicted peak VO2 at Week 16 and Year 1. Participants were assumed to be developmentally able if they had a CPX exercise assessment at any visit during study A1481131 (NCT00159913). The CPX tests were performed as close to trough plasma levels of sildenafil as possible, i.e., prior to dosing and at least 4 hours after the previous dose. If participants were able to perform the CPX test in Study A1481131 (NCT00159913), they were expected to be able to perform the exercise paradigm in the extension study (A1481156) unless their clinical condition had deteriorated and the investigator considered this was unsafe for the participant.
Time Frame: Baseline, Year 1
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Sildenafil Low/Low Dose | Sildenafil Medium/ Medium Dose | Sildenafil High/ High Dose | Placebo/ Low Dose | Placebo/ Medium Dose | Placebo/ High Dose | Placebo Non-randomized
Number analyzed (Participants) | 28 | 28 | 29 | 10 | 8 | 11 | 1
Percent | 12.79 (22.71) | 7.65 (34.57) | 5.83 (23.54) | 8.70 (25.99) | 0.20 (22.32) | -6.13 (7.46) | NA (NA) — There was no observation at Year 1 for this group

17. Secondary Outcome: Percent Change From Baseline in Time to Maximum VO2 at Year 1
Description: Exercise Tolerance Test (CPX test) was performed on developmentally able participants to determine the time to maximum VO2. Participants were assumed to be developmentally able if they had a CPX exercise assessment at any visit during study A1481131 (NCT00159913). The CPX tests were performed as close to trough plasma levels of sildenafil as possible, i.e., prior to dosing and at least 4 hours after the previous dose. If participants were able to perform the CPX test in Study A1481131 (NCT00159913), they were expected to be able to perform the exercise paradigm in the extension study (A1481156) unless their clinical condition had deteriorated and the investigator considered this was unsafe for the participant.
Time Frame: Baseline, Year 1
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Sildenafil Low/Low Dose | Sildenafil Medium/ Medium Dose | Sildenafil High/ High Dose | Placebo/ Low Dose | Placebo/ Medium Dose | Placebo/ High Dose | Placebo Non-randomized
Number analyzed (Participants) | 28 | 28 | 29 | 10 | 8 | 11 | 1
Percent | 25.47 (35.67) | 13.08 (33.42) | 7.70 (33.01) | 21.17 (57.25) | 36.68 (101.65) | -9.64 (15.21) | NA (NA) — There is no observation

18. Secondary Outcome: Percent Change From Baseline in Respiratory Exchange Ratio at Year 1
Description: This is the ratio of carbon dioxide (CO2) produced to O2 consumed [VCO2/VO2]. Exercise Tolerance Test was performed on developmentally able participants to determine the respiratory exchange ratio on week 16 and Year 1. Participants were assumed to be developmentally able if they had a CPX exercise assessment at any visit during study A1481131 (NCT00159913).
Time Frame: Baseline, Year 1
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Sildenafil Low/Low Dose | Sildenafil Medium/ Medium Dose | Sildenafil High/ High Dose | Placebo/ Low Dose | Placebo/ Medium Dose | Placebo/ High Dose | Placebo Non-randomized
Number analyzed (Participants) | 28 | 28 | 29 | 10 | 8 | 11 | 1
Percent | 2.15 (8.73) | 5.63 (13.37) | 0.68 (11.50) | -3.69 (7.24) | 0.27 (11.04) | 10.75 (17.76) | NA (NA) — There is no observation

19. Secondary Outcome: Percent Change From Start of Sildenafil in Total Ventilation (VE) to Year 1
Description: Exercise Tolerance Test (CPX test) was performed on developmentally able participants to determine the total ventilation. Participants were assumed to be developmentally able if they had a CPX exercise assessment at any visit during study A1481131 (NCT00159913). The CPX tests were performed as close to trough plasma levels of sildenafil as possible, i.e., prior to dosing and at least 4 hours after the previous dose. If participants were able to perform the CPX test in Study A1481131 (NCT00159913), they were expected to be able to perform the exercise paradigm in the extension study (A1481156) unless their clinical condition had deteriorated and the investigator considered this was unsafe for the participant.
Time Frame: Year 1
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Sildenafil Low Dose | Sildenafil Medium Dose | Sildenafil High Dose
Number analyzed (Participants) | 38 | 36 | 40
Percent | 14.29 (21.38) | 12.38 (32.64) | 11.80 (19.79)

20. Secondary Outcome: Percentage Change From Baseline in End Tidal Oxygen (O2) at Year 1.
Description: Exercise Tolerance Test (CPX test) was performed on developmentally able participants to measure the End Tidal O2 at Year 1. Participants were assumed to be developmentally able if they had a CPX exercise assessment at any visit during study A1481131 (NCT00159913). The CPX tests were performed as close to trough plasma levels of sildenafil as possible, i.e., prior to dosing and at least 4 hours after the previous dose. If participants were able to perform the CPX test in Study A1481131 (NCT00159913), they were expected to be able to perform the exercise paradigm in the extension study (A1481156) unless their clinical condition had deteriorated and the investigator considered this was unsafe for the participant.
Time Frame: Baseline, Year 1
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Sildenafil Low Dose | Sildenafil Medium Dose | Sildenafil High Dose
Number analyzed (Participants) | 25 | 22 | 24
Percent | 0.59 (3.79) | -0.52 (3.55) | 0.08 (3.68)

21. Secondary Outcome: Percentage Change From Baseline in End Tidal Carbon Dioxide (CO2) at Year 1.
Description: Exercise Tolerance Test (CPX test) was performed on developmentally able participants to measure the End Tidal CO2 at Year 1. Participants were assumed to be developmentally able if they had a CPX exercise assessment at any visit during study A1481131 (NCT00159913). The CPX tests were performed as close to trough plasma levels of sildenafil as possible, i.e., prior to dosing and at least 4 hours after the previous dose. If participants were able to perform the CPX test in Study A1481131 (NCT00159913), they were expected to be able to perform the exercise paradigm in the extension study (A1481156) unless their clinical condition had deteriorated and the investigator considered this was unsafe for the participant.
Time Frame: Baseline, Year 1
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Sildenafil Low Dose | Sildenafil Medium Dose | Sildenafil High Dose
Number analyzed (Participants) | 24 | 20 | 22
Percent | 7.83 (16.35) | 7.68 (18.74) | 13.16 (31.38)

22. Secondary Outcome: Percentage Change From Baseline in Anaerobic Threshold at Year 1.
Description: Exercise Tolerance Test (CPX test) was performed on developmentally able participants to measure the anaerobic threshold at Week 16 and Year 1. Participants were assumed to be developmentally able if they had a CPX exercise assessment at any visit during study A1481131 (NCT00159913). The CPX tests were performed as close to trough plasma levels of sildenafil as possible, i.e., prior to dosing and at least 4 hours after the previous dose. If participants were able to perform the CPX test in Study A1481131 (NCT00159913), they were expected to be able to perform the exercise paradigm in the extension study (A1481156) unless their clinical condition had deteriorated and the investigator considered this was unsafe for the participant.
Time Frame: Baseline, Year 1
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Sildenafil Low/Low Dose | Sildenafil Medium/ Medium Dose | Sildenafil High/ High Dose | Placebo/ Low Dose | Placebo/ Medium Dose | Placebo/ High Dose | Placebo Non-randomized
Number analyzed (Participants) | 26 | 27 | 28 | 10 | 7 | 10 | 1
Percent | -1.22 (23.06) | 1.99 (29.54) | 3.28 (29.36) | 7.23 (12.31) | -3.59 (28.29) | 8.96 (32.55) | NA (NA) — There was no observation at year 1 for this group

23. Secondary Outcome: Summary of Shift in Changes From Start of Sildenafil in World Health Organization Pulmonary Hypertension (WHO PH) Functional Class by A1481156 Treatment Group at Year 1.
Description: The WHO PH functional classification was as follows: Class I : Participants with PH but without resulting limitation of physical activity. Class II : Participants with PH resulting in slight limitation of physical activity. Class III : Participants with PH resulting in marked limitation of physical activity. Class IV : Participants with PH with inability to carry out any physical activity without symptoms. Changes from baseline in functional class were summarized at Years 1, 2, 3, and 4. Numbers of participants improving by 3 classes, improving by 2 classes, improving by 1 class, not changing, worsening by 1 class, worsening by 2 classes or worsening by 3 classes from A1481131 baseline at Years 1, 2, 3 and 4 were evaluated.
Time Frame: Baseline, Year 1
Population: An ITT population included all randomly assigned participants who took at least 1 dose of study medication in base study and certain analyses were conducted at pre-specified time points: 1, 2 years and 3, 4 and 5 years (where data quantity allowed) from A1481131 (NCT00159913) baseline.
Measure: Number; unit: Participants
Arm/Group | Sildenafil Low Dose | Sildenafil Medium Dose | Sildenafil High Dose
Number analyzed (Participants) | 55 | 74 | 100
Participants
  Improved by 3 Classes | 0 | 0 | 0
  Improved by 2 Classes | 1 | 0 | 1
  Improved by 1 Class | 13 | 15 | 19
  No change | 30 | 48 | 64
  Worsened by 1 Class | 4 | 6 | 3
  Worsened by 2 Classes | 1 | 0 | 0
  Worsened by 3 Classes | 0 | 0 | 0
  Discontinued | 5 | 4 | 10
  Died | 0 | 0 | 1
  Missing | 1 | 1 | 2

24. Secondary Outcome: Summary of Shift in Changes From Start of Sildenafil in WHO PH Functional Class by A1481156 Treatment Group at Year 2.
Description: The WHO PH functional classification was as follows: Class I : Participants with PH but without resulting limitation of physical activity. Class II : Participants with PH resulting in slight limitation of physical activity. Class III : Participants with PH resulting in marked limitation of physical activity. Class IV : Participants with PH with inability to carry out any physical activity without symptoms. Changes from baseline in functional class were summarised at Years 1, 2, 3, and 4. Numbers of participants improving by 3 classes, improving by 2 classes, improving by 1 class, not changing, worsening by 1 class, worsening by 2 classes or worsening by 3 classes from A1481131 baseline at Years 1, 2, 3 and 4 were evaluated.
Time Frame: Baseline, Year 2
Population: as for outcome 23
Measure: Number; unit: Participants
Arm/Group | Sildenafil Low Dose | Sildenafil Medium Dose | Sildenafil High Dose
Number analyzed (Participants) | 55 | 74 | 100
Participants
  Improved by 3 Classes | 0 | 0 | 0
  Improved by 2 Classes | 0 | 1 | 1
  Improved by 1 Class | 11 | 11 | 16
  No change | 28 | 47 | 55
  Worsened by 1 Class | 3 | 2 | 5
  Worsened by 2 Classes | 0 | 0 | 0
  Worsened by 3 Classes | 0 | 0 | 0
  Discontinued | 9 | 9 | 16
  Died | 1 | 2 | 5
  Missing | 3 | 2 | 2

25. Secondary Outcome: Summary of Shift in Changes From Start of Sildenafil in WHO PH Functional Class by A1481156 Treatment Group at Year 3.
Description: The WHO PH functional classification was as follows: Class I : Participants with PH but without resulting limitation of physical activity. Class II : Participants with PH resulting in slight limitation of physical activity. Class III : Participants with PH resulting in marked limitation of physical activity. Class IV : Participants with PH with inability to carry out any physical activity without symptoms. Changes from baseline in functional class were summarised at Years 1, 2, 3, and 4. Numbers of participants improving by 3 classes, improving by 2 classes, improving by 1 class, not changing, worsening by 1 class, worsening by 2 classes or worsening by 3 classes from A1481131 (NCT00159913) baseline at Years 1, 2, 3 and 4 were evaluated.
Time Frame: Baseline, Year 3
Population: An ITT population included all randomized participants who took at least 1 dose of study medication in base study and certain analyses were conducted at pre-specified time points: 1, 2 years and 3, 4 and 5 years (where data quantity allowed) from A1481131 (NCT00159913) baseline.
Measure: Number; unit: Participants
Arm/Group | Sildenafil Low Dose | Sildenafil Medium Dose | Sildenafil High Dose
Number analyzed (Participants) | 55 | 74 | 100
Participants
  Improved by 3 Classes | 0 | 0 | 0
  Improved by 2 Classes | 1 | 0 | 1
  Improved by 1 Class | 11 | 16 | 17
  No change | 21 | 36 | 44
  Worsened by 1 Class | 3 | 3 | 5
  Worsened by 2 Classes | 1 | 0 | 1
  Worsened by 3 Classes | 0 | 0 | 0
  Discontinued | 14 | 13 | 19
  Died | 2 | 3 | 9
  Missing | 2 | 3 | 4

26. Secondary Outcome: Summary of Shift in Changes From Start of Sildenafil in WHO PH Functional Class by A1481156 Treatment Group at Year 4.
Description: as for outcome 24
Time Frame: Baseline, Year 4
Population: as for outcome 23
Measure: Number; unit: Participants
Arm/Group | Sildenafil Low Dose | Sildenafil Medium Dose | Sildenafil High Dose
Number analyzed (Participants) | 55 | 74 | 100
Participants
  Improved by 3 Classes | 0 | 0 | 0
  Improved by 2 Classes | 0 | 0 | 2
  Improved by 1 Class | 13 | 14 | 16
  No change | 15 | 29 | 41
  Worsened by 1 Class | 6 | 4 | 5
  Worsened by 2 Classes | 1 | 2 | 1
  Worsened by 3 Classes | 0 | 0 | 0
  Discontinued | 15 | 18 | 20
  Died | 2 | 5 | 13
  Missing | 3 | 2 | 2

27. Secondary Outcome: Additions From Baseline in Background Therapy up to the End of Study
Description: This was defined as an addition or discontinuation in the class(es) of drugs used as background medication (e.g., anticoagulants, oxygen, diuretics, calcium channel blockers, and digoxin) compared to baseline of Study A1481131 (NCT00159913).
Time Frame: Up to the end of study
Population: as for outcome 23
Measure: Number; unit: Participants
Arm/Group | Sildenafil Low/Low Dose | Sildenafil Medium/ Medium Dose | Sildenafil High/ High Dose | Placebo/ Low Dose | Placebo/ Medium Dose | Placebo/ High Dose | Placebo Non-randomized
Number analyzed (Participants) | 42 | 55 | 77 | 13 | 19 | 23 | 5
Participants
  All Classes (N = 18, 26, 43, 7, 8, 14, 4) | 6 | 5 | 11 | 2 | 1 | 2 | 1
  At least one class (N = 42, 55, 77, 13, 19, 23, 5) | 13 | 13 | 23 | 3 | 5 | 2 | 1

28. Secondary Outcome: Change From Baseline in Child Health Questionnaire-Parent Form (CHQ-PF28) as Assessed by the Psychosocial Scale at Year 1.
Description: CHQ: 50-item, 15 subscale parent or legal guardian assessed instrument of child's physical, emotional, social well-being, and relative burden of disease on the parents; rated on Likert-type scale: range 0 to 100; higher scores indicate a more positive health status. Global indicators for Physical Health and Psychosocial Health are weighted composites derived from subscale items using scoring algorithms (transformed scores); range 0 to 100: higher scores indicate more positive health status.
Time Frame: Baseline, Year 1
Population: ITT population included all randomized participants who took at least 1 dose of study drug in base study; certain analyses were conducted at pre-specified time points: 1, 2 years and 3, 4, 5 years (where data quantity allowed) from A1481131 (NCT00159913) baseline. Participants >= 5 years at baseline with questionnaire translated were included.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sildenafil Low/Low Dose | Sildenafil Medium/ Medium Dose | Sildenafil High/ High Dose | Placebo/ Low Dose | Placebo/ Medium Dose | Placebo/ High Dose | Placebo Non-randomized
Number analyzed (Participants) | 34 | 30 | 45 | 11 | 14 | 15 | 1
Units on a scale | 5.63 (7.70) | 3.92 (10.25) | 3.48 (12.55) | 13.74 (12.42) | 5.30 (9.30) | 4.27 (12.19) | NA (NA) — There was no observation at year 1 this group

29. Secondary Outcome: Change From Baseline in Child Health Questionnaire-Parent Form (CHQ-PF28) as Assessed by the Physical Scale at Year 1.
Description: as for outcome 28
Time Frame: Baseline, Year 1
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sildenafil Low/Low Dose | Sildenafil Medium/ Medium Dose | Sildenafil High/ High Dose | Placebo/ Low Dose | Placebo/ Medium Dose | Placebo/ High Dose | Placebo Non-randomized
Number analyzed (Participants) | 34 | 30 | 45 | 11 | 14 | 15 | 1
Units on a scale | 14.29 (11.06) | 9.34 (13.45) | 5.91 (10.17) | 8.51 (13.27) | 9.86 (17.93) | 4.64 (12.03) | NA (NA) — There was no observation at year 1 for placebo/non-randomized

30. Secondary Outcome: Participant (Parent) Global Assessment at Year 1
Description: The participant (parent) global assessment of disease severity was assessed at Year 1 in this extension study. The number and percentage of participants markedly improved, moderately improved, mild improvement, no change, slightly worse, moderately worse, markedly worse were evaluated. Participants who withdrew from study treatment after at least 10 weeks of treatment were requested to perform the global assessments.
Time Frame: Year 1
Population: as for outcome 23
Measure: Number; unit: Participants
Arm/Group | Sildenafil Low Dose | Sildenafil Medium Dose | Sildenafil High Dose
Number analyzed (Participants) | 55 | 74 | 100
Participants
  Markedly Improved | 9 | 14 | 21
  Moderately Improved | 13 | 27 | 26
  Mild Improvement | 12 | 15 | 15
  No Change | 13 | 6 | 21
  Slightly Worse | 1 | 2 | 0
  Moderately Worse | 0 | 1 | 0
  Markedly Worse | 0 | 0 | 0
  Discontinued | 5 | 4 | 10
  Died | 0 | 0 | 1
  Missing | 2 | 5 | 6

31. Secondary Outcome: Physician Global Assessment at Year 1
Description: The physician global assessment of disease severity was assessed at Year 1 in this extension study. The number and percentage of participants with markedly improved, moderately improved, mild improvement, no change, slightly worse, moderately worse, markedly worse were evaluated. Participants who withdrew from study treatment after at least 10 weeks of treatment were requested to perform the global assessments.
Time Frame: Year 1
Population: as for outcome 23
Measure: Number; unit: Participants
Arm/Group | Sildenafil Low Dose | Sildenafil Medium Dose | Sildenafil High Dose
Number analyzed (Participants) | 55 | 74 | 100
Participants
  Markedly Improved | 6 | 6 | 6
  Moderately Improved | 8 | 18 | 27
  Mild Improvement | 19 | 26 | 37
  No Change | 15 | 16 | 17
  Slightly Worse | 1 | 1 | 0
  Moderately Worse | 0 | 1 | 0
  Markedly Worse | 0 | 0 | 0
  Discontinued | 5 | 4 | 10
  Died | 0 | 0 | 1
  Missing | 1 | 2 | 2

ADVERSE EVENTS:
Time Frame: Up to Follow-Up visit (30 to 40 days after study completion or treatment discontinuation)
Description: The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Sildenafil Low Dose | Sildenafil Medium Dose | Sildenafil High Dose
Serious Adverse Events (participants affected / at risk) | 14/55 | 37/74 | 48/100
Other Adverse Events (participants affected / at risk) | 51/55 | 70/74 | 87/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sildenafil Low Dose (N=55) | Sildenafil Medium Dose (N=74) | Sildenafil High Dose (N=100)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Polycythaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 2 | 2 | 6
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 2
Cyanosis (Cardiac disorders) | 1 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Right ventricular failure (Cardiac disorders) | 2 | 3 | 3
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Tachycardia paroxysmal (Cardiac disorders) | 0 | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 2
Cystic fibrosis (Congenital, familial and genetic disorders) | 0 | 1 | 0
Eisenmenger's syndrome (Congenital, familial and genetic disorders) | 0 | 1 | 0
Hip dysplasia (Congenital, familial and genetic disorders) | 1 | 1 | 0
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 0 | 1
Corneal oedema (Eye disorders) | 0 | 0 | 1
Keratoconus (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Chest pain (General disorders) | 3 | 0 | 2
Disease progression (General disorders) | 0 | 1 | 0
Gait disturbance (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 3
Acute tonsillitis (Infections and infestations) | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Brain abscess (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 3
Bronchopneumonia (Infections and infestations) | 1 | 1 | 3
Cellulitis (Infections and infestations) | 0 | 1 | 0
Dengue fever (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 3 | 3
Gastroenteritis salmonella (Infections and infestations) | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 1
Gingivitis (Infections and infestations) | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 7 | 10
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 6
Urinary tract infection (Infections and infestations) | 0 | 0 | 3
Viral infection (Infections and infestations) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Exposure via father (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Catheterisation cardiac (Investigations) | 0 | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 1
Pulmonary arterial pressure increased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 1 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 2 | 2 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Anorexia nervosa (Psychiatric disorders) | 1 | 0 | 0
Enuresis (Renal and urinary disorders) | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 7
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 5
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Cardiac operation (Surgical and medical procedures) | 0 | 1 | 0
Central venous catheterisation (Surgical and medical procedures) | 0 | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sildenafil Low Dose (N=55) | Sildenafil Medium Dose (N=74) | Sildenafil High Dose (N=100)
Hypothyroidism (Endocrine disorders) | 0 | 4 | 0
Conjunctival hyperaemia (Eye disorders) | 3 | 5 | 6
Conjunctivitis (Eye disorders) | 1 | 3 | 9
Conjunctivitis allergic (Eye disorders) | 0 | 4 | 3
Retinal vascular disorder (Eye disorders) | 1 | 4 | 6
Visual acuity reduced (Eye disorders) | 2 | 4 | 5
Visual impairment (Eye disorders) | 3 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 4 | 4 | 13
Abdominal pain upper (Gastrointestinal disorders) | 3 | 5 | 9
Dental caries (Gastrointestinal disorders) | 6 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 10 | 11 | 16
Dyspepsia (Gastrointestinal disorders) | 3 | 6 | 5
Gastritis (Gastrointestinal disorders) | 2 | 4 | 5
Nausea (Gastrointestinal disorders) | 2 | 5 | 12
Vomiting (Gastrointestinal disorders) | 14 | 13 | 24
Chest pain (General disorders) | 5 | 4 | 12
Fatigue (General disorders) | 4 | 8 | 7
Pyrexia (General disorders) | 7 | 16 | 16
Bronchitis (Infections and infestations) | 10 | 16 | 16
Bronchopneumonia (Infections and infestations) | 0 | 4 | 2
Ear infection (Infections and infestations) | 3 | 8 | 4
Gastroenteritis (Infections and infestations) | 4 | 3 | 7
Influenza (Infections and infestations) | 10 | 6 | 12
Laryngitis (Infections and infestations) | 5 | 1 | 4
Nasopharyngitis (Infections and infestations) | 15 | 11 | 17
Otitis media (Infections and infestations) | 2 | 4 | 4
Pharyngitis (Infections and infestations) | 16 | 13 | 13
Pharyngitis streptococcal (Infections and infestations) | 3 | 3 | 2
Pneumonia (Infections and infestations) | 2 | 4 | 0
Respiratory tract infection (Infections and infestations) | 2 | 4 | 5
Rhinitis (Infections and infestations) | 6 | 10 | 7
Sinusitis (Infections and infestations) | 2 | 3 | 8
Tonsillitis (Infections and infestations) | 9 | 6 | 13
Upper respiratory tract infection (Infections and infestations) | 9 | 22 | 37
Urinary tract infection (Infections and infestations) | 3 | 2 | 6
Varicella (Infections and infestations) | 3 | 3 | 4
Blood pressure diastolic decreased (Investigations) | 3 | 3 | 4
Weight decreased (Investigations) | 3 | 2 | 3
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 3 | 2
Dizziness (Nervous system disorders) | 7 | 4 | 10
Headache (Nervous system disorders) | 18 | 18 | 26
Syncope (Nervous system disorders) | 5 | 7 | 5
Insomnia (Psychiatric disorders) | 3 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 14 | 17
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 12 | 9
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 5
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 9
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.